CLINICAL TRIAL: NCT00195403
Title: A Drug Use Investigation of Enbrel for Post-Marketing Surveillance
Brief Title: A Drug Use Investigation of ENBREL for Post-marketing Surveillance (PMS) for RA and PsA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101575
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 25mg Injection, 2 times/week

SUMMARY:
The objective of this investigation is to identify the following problems and questions with respect to the safety and efficacy of Enbrel during the post-marketing period as required by Korea Food and Drug Administration (KFDA)'s regulation.

1. Unknown adverse reactions, especially serious adverse reactions
2. Incidences of adverse reactions under routine drug uses
3. Factors that may affect the safety of the drug
4. Factors that may affect the efficacy of the drug

This investigation spanned 3 different studies, 0881A-101575 (alias B1801105) NCT00195403, 0881A-102018 (alias B1801112) NCT00195416 and 0881A-102212 (alias B1801113). All studies have been combined into this record.

ELIGIBILITY:
Inclusion Criteria

Rheumatoid Arthritis

* Adults: Treatment of active rheumatoid arthritis (RA) in adults when the response to disease-modifying antirhematic drugs (DMARDs), including MTX, has been inadequate
* Children: Treatment of active polyarticular-course chronic active rheumatoid arthritis in children aged 4 to 17 years who have had an inadequate response to, or whom have proved intolerant of, MTX

Psoriatic Arthritis

- Active and progressive psoriatic arthritis (PsA) in adults who do not respond adequately to previous DMARDs

Exclusion Criteria

* Patients to whom Enbrel is contraindicated as per the local labeling
* Patients with known hypersensitivity to Enbrel or any component of the product
* Patients with sepsis or risk of sepsis
* Patients with active infections including chronic or localized infections such as tuberculosis. (Treatment of Enbrel should not be initiated.)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic, secondary and tertiary medical centers
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2004-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- South Korea (2):
  - Kyunggi-do
  - Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results for three unique protocols 0881A-101575 (NCT00195403), 0881A-102018 (NCT00195416), and 0881A-102212 (protocol not registered) were summarized in a single clinical study report.
Pre-assignment Details: Total of 1016 case report forms were retrieved, of these 2 were double registered. Out of 1014 participants, 16 were enrolled prior to the agreement date of the study and therefore excluded from the safety analysis population (998). Three participants had missing efficacy assessments (efficacy population = 995).
Groups:
- Etanercept: Participants who had rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis and received etanercept subcutaneously as per local medical practitioner's discretion were observed up to 6 years. The recommended etanercept dose is 25 milligram (mg) subcutaneously twice weekly or 50 mg subcutaneously once weekly.
Period: Overall Study
Arm/Group | Etanercept
Started | 1014
Completed | 1014
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least (>=) 1 dose of study medication and had the safety assessment through appropriate follow-up.
Arm/Group | Etanercept
Number analyzed (Participants) | 998
Age Continuous [Mean (Standard Deviation); unit: years] | 40.21 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 465
  Male | 533
Primary diagnosis [Number; unit: participants]
  Ankylosing Spondylitis | 520
  Rheumatoid Arthritis | 475
  Psoriatic Arthritis | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an AE, without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a serious AE (SAE): death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Unexpected AEs were reported as yes or no at the investigator's determination based on current country product label.
Time Frame: Baseline up to Day 832
Population: Safety population included all participants who received >= 1 dose of study medication and had the safety assessment through appropriate follow-up.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 998
participants
  Any adverse event | 142
  Serious adverse event | 3
  Unexpected adverse event | 27

2. Primary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Disease Status at Month 3
Description: PGA of disease activity was measured on a 0 to 10 centimeter (cm) Visual Analog Scale (VAS), with 0 cm = no disease activity and 10 cm = worst disease activity possible.
Time Frame: Baseline, Month 3
Population: Efficacy population included all participants who received >=1 dose of study medication and had the efficacy assessment within 14 days after the final administration.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 995
cm
  Baseline | 7.49 (1.30)
  Change at Month 3 | -4.34 (1.86)
Statistical Analysis 1: Comparison: Etanercept; Change from baseline in PGA at Month 3 was evaluated using paired t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Number of Joints With Tenderness, Pain, Limitation of Motion or Swelling at Month 3 and 9
Description: Assessment of 68 joints: joints classified as either tender or not tender, pain or no pain, with limitation of motion or no limitation of motion, swollen or not swollen. An increase from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Month 3, 9
Population: Efficacy population included all participants who received >=1 dose of study medication and had the efficacy assessment within 14 days after the final administration. 'N' (number of participants analyzed) = participants who were evaluable for this measure. Data for Month 9 was not analyzed because there were not enough participants for analysis.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Etanercept
Number analyzed (Participants) | 430
joints
  Baseline | 17.42 (11.37)
  Change at Month 3 | -12.67 (9.91)
Statistical Analysis 1: Comparison: Etanercept; Change from baseline in number of joints with tenderness, pain, and limitation of motion or swelling at Month 3 were evaluated using paired t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Description: All adverse events which occurred in the participants collected during the study period were included in reports regardless of their causal relationship with the study drug.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 3/998
Other Adverse Events (participants affected / at risk) | 142/998
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=998)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Herpes zoster (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=998)
Itching (Skin and subcutaneous tissue disorders) | 36
Rash (Skin and subcutaneous tissue disorders) | 9
Urticaria (Skin and subcutaneous tissue disorders) | 1
Macular rash (Skin and subcutaneous tissue disorders) | 1
Verruca vulgatis (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Burn (Skin and subcutaneous tissue disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Injection site itching (General disorders) | 12
Injection site erythema (General disorders) | 7
Injection site reaction (General disorders) | 3
Injection site edema (General disorders) | 3
Injection site pain (General disorders) | 3
Cellulitis (General disorders) | 1
Injection site burning sensation (General disorders) | 1
Headache (General disorders) | 7
Edema (General disorders) | 6
Facial flushing (General disorders) | 3
Fever (General disorders) | 3
Chest pain (General disorders) | 2
Facial edema (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5
Increased Serum Glutamic Pyruvate Transaminase (Hepatobiliary disorders) | 4
Increased Serum Glutamic-oxaloacetic Transminase (Hepatobiliary disorders) | 3
Hepatotoxicity (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Infection, aggravated (Infections and infestations) | 1
Tuberculosis, bones and joints (Infections and infestations) | 1
Abscess, pulmonary (Infections and infestations) | 1
Ear discharge (Infections and infestations) | 1
Shock, septic (Infections and infestations) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thirst (Metabolism and nutrition disorders) | 1
Weight decrease (Metabolism and nutrition disorders) | 1
Weight increase (Metabolism and nutrition disorders) | 1
Auto-antibody response (General disorders) | 1
Uveitis (Eye disorders) | 2
Xerophthalmia (Eye disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Blood pressure high (General disorders) | 1
Lymph nodes enlarged (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Azotemia (Renal and urinary disorders) | 1
Palpitation (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.